CLINICAL TRIAL: NCT05367596
Title: OPTIMIzing muScle Preservation in paTients wIth Cirrhosis
Acronym: OPTIMISTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Winston Dunn, M.D., Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00148145
Record Dates: First submitted 2022-05-02; First posted 2022-05-10 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Compensated Cirrhosis; Sarcopenia
MeSH Terms: conditions — Obesity; Sarcopenia | interventions — Exercise; Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Energy Restriction (CER) (Experimental): Continuous energy restriction (CER; 1,200-1,500 kcal/day). Participants in both groups will have a daily late-evening snack and participate in remotely supervised exercises.
  Interventions: Behavioral: Continuous Energy Restriction (CER); Behavioral: Group Health Education Sessions; Behavioral: Late Evening Snack; Behavioral: Physical activity; Behavioral: Self-monitoring; Behavioral: Remotely Supervised Exercise Sessions
- Alternate-Day Moderate Fasting (ADMF). (Experimental): Alternate-Day Moderate Fasting (ADMF). Participants in both groups will have a daily late-evening snack and participate in remotely supervised exercises.
  Interventions: Behavioral: Alternate Day Modified Fasting (ADMF); Behavioral: Group Health Education Sessions; Behavioral: Late Evening Snack; Behavioral: Physical activity; Behavioral: Self-monitoring; Behavioral: Remotely Supervised Exercise Sessions

INTERVENTIONS:
Behavioral: Continuous Energy Restriction (CER) — Energy intake will be prescribed at approximately 1,200-1,500 kcal/day with high protein. The diet will consist of low-calorie shakes provided by the study, as well as commercially available portion-controlled entrées, fruits/vegetables, and low energy-density foods available in grocery stores.
  Arms: Continuous Energy Restriction (CER)
Behavioral: Alternate Day Modified Fasting (ADMF) — Enhanced Care participants will have an alternate between three days of very-low energy intake (VLED; approximately 600-800 kcal/d) and four days of healthy eating (HE) each week. On HE days, participants will consume foods ad libitum for satiety.
  Arms: Alternate-Day Moderate Fasting (ADMF).
Behavioral: Group Health Education Sessions — Using video conferencing, all participants will attend weekly approximately 45-60 minutes group health education sessions led by a registered dietitian. The session will deliver a comprehensive nutritional and lifestyle change program to promote lifestyle changes and improve compliance.
Behavioral: Late Evening Snack — The participants will have a late evening snack with a protein supplement.
Behavioral: Physical activity — All participants will be prescribed moderate-intensity aerobic activities that do not require access to specialized exercise facilities.
Behavioral: Self-monitoring — Weekly data related to adherence, food intake, physical activity, weight measurement, and nonserious adverse events will be self-reported via a REDCap survey. Participants will also be provided with a wireless activity tracker to measure total physical activity and intensity of activity objectively. These data will be used to counsel participants in addition to providing valuable feasibility data.
Behavioral: Remotely Supervised Exercise Sessions — Sessions of 45 minutes duration will be delivered via video conferencing 2-3 times per week.

SUMMARY:
Patients with obesity and cirrhosis benefit from weight loss but are prone to sarcopenia (loss of muscle mass, strength, and function).

This study proposes to test a specialized weight loss program Alternative-day Modified Fasting (ADMF) designed to promote weight loss and preserve skeletal muscle mass, strength, and function in patients with both Child-Pugh (CP) class A cirrhosis and obesity. This study will compare the effectiveness of the ADMF to Continuous Energy Restriction (CER) for 24-weeks. Both arms will receive a high-protein, high-BCAA diet, a late-night snack, supervised aerobic and resistance exercise, increased physical activity through self-monitoring, and group behavioral counseling.

The primary aim of this trial is to evaluate the feasibility and acceptability of ADMF and CER for 6 months in patients with cirrhosis and obesity. The secondary aim is to compare changes in body composition in both diets.

DETAILED DESCRIPTION:
Patients with both cirrhosis and obesity benefit from weight loss, though patients with cirrhosis are prone to sarcopenia due to accelerated rates of protein turnover, and weight loss typically involves 20-30% of weight loss from lean mass. Prior research indicates that increased intake of high-quality protein, reduced fasting duration, and regular physical activity (particularly resistance training) can improve body composition in patients with cirrhosis. However, weight loss programming specifically tailored to retain lean mass in patients with cirrhosis has not been thoroughly investigated. Further, preliminary data suggests that alternate-day modified fasting, a form of intermittent fasting, may promote lean mass retention during weight loss. Here, this study will compare a weight loss program in patients with both Child-Pugh Class A cirrhosis and obesity using either a standard low-calorie diet (1,200 - 1,500 kcal/day) or alternate day modified fasting featuring a very-low-calorie diet 2-3 days per week for feasibility, satisfaction, and changes in body composition. Both groups will receive a behavioral weight loss program featuring portion-controlled meals and supervised group exercise.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age. Per the NIH Policy NOT-OD-18-116, we will include adults ≥ 65 yrs.
* Subjects have a BMI of 30-45. Body mass index (BMI) of 25 to 45 kg/m2. Individuals with a BMI< 25 kg/m2 are not overweight, and individuals with a BMI >45 kg/m2 require more aggressive weight-loss interventions such as bariatric surgery.
* Subjects has a diagnosis of cirrhosis based on any of the following methods

  * Liver Biopsy is consistent with stage IV fibrosis according to the NASH Clinical Research Network (CRN) scoring system.
  * Fibroscan Liver Stiffness >14kpa
  * Endoscopy or imaging finding of varices

Exclusion Criteria:

* Child-Pugh (CP) score currently > 6 (i.e., CP Class B/C cirrhosis).
* History of ascites.
* History of portal system encephalopathy.
* Prior history of liver cancer.
* Prior history of non-melanoma skin cancer within the last five years
* Hepatitis C Virus (HCV) patients who have not undergone sustained virological response (SVR).
* Hepatitis B Virus (HBV) Patients who have not received antiviral treatment.
* Patients with diabetes currently on insulin and or sulfonylureas.
* Active alcohol use >7 drinks per week in the past six months.
* Suspected eating disorders based on Eating Attitudes Test (EAT-26) and The Binge Eating Scale (BES):
* Unable to participate in moderate-intensity PA, e.g., brisk walking
* Participation in a structured weight loss program in the previous six mos.
* Not weight stable (5%) for three months prior to intake.
* Unwilling to be randomized.
* Pregnancy during the previous six mos., currently lactating, or planned pregnancy in the following six mos
* Current use of antipsychotics, untreated depression, or other psychiatric illnesses would preclude weight management participation.
* Adherence to specialized diets that would make it difficult or impossible to follow the guidelines for intervention.
* Evidence of eating disorder or binge eating (as assessed by the Eating Attitudes Test and or Binge Eating Scale.)
* Do not have access to a wireless equipment necessary for remotely delivered group and exercise classes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Compare changes in body composition in both diets | Baseline, 12 weeks and 24 weeks.
  The primary outcome is the percent of weight lost as fat-free mass at 24 weeks. Body weight and body composition (as assessed by dual x-ray absorptiometry) will be measured at baseline, week 12, and post-intervention. Percent weight loss from fat-free mass will be calculated as [Δ fat-free mass / Δ weight loss] for all participants who lose at least 3% of initial body weight. If >70% of participants lose at least 80% of weight from fat mass (or no more than 20% of weight loss coming from lean mass) we will proceed to testing this intervention in an adequately powered trial.

SECONDARY OUTCOMES:
Frailty, Subjective | Baseline, 12 weeks and 24 weeks.
  Karnofsky Performance Status (KPS). The KPS allows patients to be classified as to their functional impairment. This can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. The lower the KPS, the worse the survival for most serious illnesses.
Frailty, Objective | Baseline, 12 weeks and 24 weeks.
  The Liver Frailty Index (LFI), composed of 3 performance-based tests (grip strength, chair stands, and balance), is a tool specifically developed in patients with cirrhosis to objectively measure physical function, a critical determinant of health outcomes.
Health Related Quality of Life | Baseline, 12 weeks and 24 weeks.
  Health-related quality of life (HRQOL) is a multi-dimensional concept commonly used to examine the impact of health status on quality of life. HRQOL is often measured by four core questions that asked about general health status and number of unhealthy days.

CONTACTS AND LOCATIONS:
Overall Officials: Winston Dunn, MD, Principal Investigator — KUMC; Felicia Felicia Steger, PhD, Principal Investigator — KUMC
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dunn W, Herrmann SD, Montgomery RN, Hastert M, Honas JJ, Rachman J, Donnelly JE, Steger FL. Optimizing muscle preservation during weight loss in patients with cirrhosis: A pilot study comparing continuous energy restriction to alternate-day modified fasting for weight loss in patients with obesity and non-alcoholic cirrhosis of the liver. Obes Sci Pract. 2024 Oct 24;10(5):e70016. doi: 10.1002/osp4.70016. eCollection 2024 Oct. PMID 39450267